CLINICAL TRIAL: NCT04148521
Title: A Virtual Navigation Intervention to Reduce Behavioral Health Admissions From Rural Emergency Departments (VIBRANT)
Brief Title: A Virtual Navigation Intervention to Reduce Behavioral Health Admissions From Rural Emergency Departments
Acronym: VIBRANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: The Duke Endowment (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00081746; 13952 (Other: Atrium Health); Pro00038573 (Other: Atrium Health)
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Results first posted 2022-04-12 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-02

CONDITIONS: Depression; Anxiety; Substance Use Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Health - Virtual Patient Navigation (Experimental): All patients who meet eligibility criteria at sites where the virtual patient navigation behavioral health program is offered will be considered exposed to the intervention.
  Interventions: Behavioral: Behavioral Health - Virtual Patient Navigation
- Usual care Behavioral Health (No Intervention): All patients who meet eligibility criteria at sites where the virtual patient navigator behavioral health program is not offered will be considered exposed to usual care.

INTERVENTIONS:
Behavioral: Behavioral Health - Virtual Patient Navigation — Patients are identified by a clinician in the ED as needing psychiatric evaluation and a referral is made to a tele-psych provider for a virtual consult. Patients can be enrolled to the intervention arm based on a randomization scheme that randomly allocates days that navigators are available. The psychiatrist will make a recommendation to admit or discharge the patient. For patients that have a discharge recommendation on days that BH-VPN is available, patients will be offered the BH-VPN program. Enrolled patients are followed for up to 45 days. On days where the navigator is available, all patients who meet eligibility criteria will be considered exposed to the intervention.
  Arms: Behavioral Health - Virtual Patient Navigation

SUMMARY:
This research project is a pragmatic, randomized evaluation of a quality improvement initiative which seeks to evaluate the effects of standardizing the use of a BH-VPN program among patients with a telepsychiatric consult. The outcomes evaluation of this intervention has been designed to integrate with routine care and minimize frontline staff burden by deploying an evaluation in a real-world setting.

DETAILED DESCRIPTION:
Hospital admissions are common amongst those with mental illness. Significant morbidity exists for patients who are being admitted to a psychiatric hospital from the Emergency Department (ED).Additionally, commitment to a hospital setting may have adverse effects on patients psychologically, degrade relationships with therapists, and disrupt continuity of care. ED providers often decide to admit to a psychiatric hospital because of limited availability of behavioral health resources. To better enhance transitions of care for those with mental illness, Atrium Health has designed a behavioral health virtual patient navigation (BH-VPN)program that helps coordinate services and follow-up care, while facilitating the safe discharge of patients. Patients presenting to an ED that have a tele psychiatric consult who are recommended for discharge are eligible for services. The Behavioral health Service line is expanding the program to additional rural emergency departments. Using an outcomes evaluation, the investigators will inform Atrium Health on the effect of the BH-VPN program to reduce hospital admissions among patients with a tele psychiatric consult in the ED. The proposed hypothesis is that by having the BH-VPN program available in an ED, more patients will be discharged from the ED than admitted.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients must meet each of the following criteria:

* Present to an ED at participating sites
* Complete a telepsychiatric consult as captured in the electronic medical record
* Complete a telepsychiatric consult during the navigator's hours of operation
* ≥ 18 years of age at time of ED admission

Exclusion Criteria:• Patients currently enrolled in the BH-VPN program upon their index ED encounter

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1089 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Roberge, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (9):
- United States (9):
  - Atrium Health - Stanly, Albemarle, North Carolina
  - Atrium Health - Kings Mountain, Kings Mountain, North Carolina
  - Scotland Memorial Hospital, Laurinburg, North Carolina
  - Atrium Health - Lincoln, Lincolnton, North Carolina
  - Carolinas HealthCare System - Blue Ridge - Morganton, Morganton, North Carolina
  - Atrium Health - Cleveland, Shelby, North Carolina
  - Carolinas HealthCare System - Valdese, Valdese, North Carolina
  - Atrium Health - Anson, Wadesboro, North Carolina
  - Columbus Regional Hospital, Whiteville, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Behavioral Health - Virtual Patient Navigation | Usual Care Behavioral Health
Started | 534 | 555
Completed | 534 | 555
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Health - Virtual Patient Navigation | Usual Care Behavioral Health | Total
Number analyzed (Participants) | 534 | 555 | 1089
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (16.0) | 41.6 (15.9) | 41.4 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 248 | 470
  Male | 312 | 307 | 619
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 91 | 92 | 183
  White | 420 | 437 | 857
  More than one race | 16 | 18 | 34
  Unknown or Not Reported | 7 | 8 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 534 | 555 | 1089

OUTCOME MEASURES:

1. Primary Outcome: Assessing Hospital Admissions
Description: Compare the effectiveness of having the Behavioral Health - Virtual Patient Navigation (BH-VPN) program available compared to usual care, on admission rates among patients in the ED with a telepsychiatric consult
Time Frame: Up to 2 weeks from initial ED admission
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Health - Virtual Patient Navigation | Usual Care Behavioral Health
Number analyzed (Participants) | 534 | 555
Participants | 332 | 326
Statistical Analysis 1: Comparison: Behavioral Health - Virtual Patient Navigation; Test type: Superiority; p = 0.27, Mixed Models Analysis; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.90 to 1.47]

2. Secondary Outcome: 45-day Post Discharge Utilization Rate
Description: Comparing the 45-day utilization (ED, IP, OBS encounter) rate after the ED encounter between the 2 arms of the study
Time Frame: 45 days
Measure: Number; unit: participants
Arm/Group | Behavioral Health - Virtual Patient Navigation | Usual Care Behavioral Health
Number analyzed (Participants) | 534 | 555
participants | 88 | 89
Statistical Analysis 1: Comparison: Behavioral Health - Virtual Patient Navigation vs Usual Care Behavioral Health; Test type: Superiority; p = 0.83, Mixed Models Analysis; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.75 to 1.43]

3. Secondary Outcome: 45-day Post Discharge Utilization Rate With a Self-harm Diagnosis
Description: Compare the frequency of patients with any encounter with a self-harm diagnosis within 45 days of the ED visit between the 2 arms of the study
Time Frame: 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Health - Virtual Patient Navigation | Usual Care Behavioral Health
Number analyzed (Participants) | 534 | 555
Participants | 47 | 35
Statistical Analysis 1: Comparison: Behavioral Health - Virtual Patient Navigation vs Usual Care Behavioral Health; Test type: Superiority; p = 0.12, Mixed Models Analysis; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.91 to 2.26]

4. Secondary Outcome: 45-day Post Discharge ED Utilization Rate With a Behavioral Health Crisis
Description: Compare the frequency of patients who return to the ED and have a telepsychiatric consult within 45 days of their initial ED visit between the 2 arms of the study
Time Frame: 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Health - Virtual Patient Navigation | Usual Care Behavioral Health
Number analyzed (Participants) | 534 | 555
Participants | 40 | 36
Statistical Analysis 1: Comparison: Behavioral Health - Virtual Patient Navigation vs Usual Care Behavioral Health; Test type: Superiority; p = 0.51, Mixed Models Analysis; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.73 to 1.86]

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Behavioral Health - Virtual Patient Navigation | Usual Care Behavioral Health
All-Cause Mortality (participants affected / at risk) | 0/534 | 0/555
Serious Adverse Events (participants affected / at risk) | 0/534 | 0/555
Other Adverse Events (participants affected / at risk) | 0/534 | 0/555

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT04148521/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT04148521/ICF_001.pdf